CLINICAL TRIAL: NCT05606016
Title: Examining How a Facilitated Self-Sampling Intervention and Testing Navigation Intervention Influences COVID-19 Testing in Vulnerable Populations
Brief Title: Examining How a Facilitated Self-Sampling Intervention and Testing Navigation Intervention Influences COVID-19 Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Maria E Fernandez, Lorne Bain Distinguished Professorship in Public Health and Director, Center for Health Promotion and Prevention Research, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-SPH-20-1372 Embedded Study; 3UL1TR003167-03S3 (NIH)
Record Dates: First submitted 2022-08-11; First posted 2022-11-04 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: COVID-19; antigen testing; decision making; testing behaviors; vulnerable populations; social networks
MeSH Terms: conditions — COVID-19 | interventions — Troponin I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Facilitated Self-Sampling Intervention (FSSI) (Experimental): Participants in the FSSI arm will receive education on COVID-19 testing and be provided with rapid antigen tests. Participants will also receive pre and post surveys.
  Interventions: Behavioral: Facilitated Self-Sampling Intervention (FSSI)
- Testing Navigation Intervention (TNI). (Experimental): Participants in the TNI arm will receive COVID-19 testing education and be navigated to PCR testing sites. Participants will also receive pre and post surveys.
  Interventions: Behavioral: Testing Navigation Intervention (TNI).
- Control (Active Comparator): Participants in the Control Group arm will receive a CDC-designed COVID-19 testing brochures, and pre and post surveys only.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Facilitated Self-Sampling Intervention (FSSI) — CHWs will consent and enroll participants to the FSSI from the randomized PBGs. FSSI will consist of Community Health Worker (CHW) delivered education intervention about COVID-19 testing at a home visit. In addition, the participant will receive a batch of 4 rapid antigen tests which can be shared with people in the household or other close contacts if needed. The CHWs will provide low-literacy instructions for administering the tests, including print and video. The CHWs will also provide guidance if they tested positive (e.g. quarantine, notify contacts, wearing a mask). The CHWs will also be available by phone to the participants for any follow-up questions. CHW will follow-up via text and phone with the participants during the two months post intervention. In addition to the intervention, the participants will be asked to complete the pre and post test surveys. Post surveys will be administered online or over the phone two months after the initial intervention.
  Arms: Facilitated Self-Sampling Intervention (FSSI)
Behavioral: Testing Navigation Intervention (TNI). — CHWs will consent and enroll participants to the TNI from the randomized PBGs. The TNI will consist of CHW-led intervention at a home visit where they will provide low health literacy materials about how and when to conduct a COVID 19 test (including antigen and PCR) using a decision tree model and provide navigation to nearby PCR testing sites, locations to purchase antigen tests and support in accessing federal government antigen tests if not already obtained by the participant. In addition to the intervention, the participants will be asked to complete the pre and post-test surveys. Post surveys will be administered online or over the phone two months after the initial intervention.
  Arms: Testing Navigation Intervention (TNI).
Behavioral: Control — Participants in the Control arm will receive CDC-designed COVID-19 testing brochures, and pre and post surveys only.
  Arms: Control

SUMMARY:
Antigen self-testing kits are more available at this stage in the pandemic, but among vulnerable populations, use is still low and instructions for antigen testing are not typically designed for low health literacy populations. Studies are needed to explore access and use of antigen tests among vulnerable populations and examine if low-health-literacy-designed interventions improve COVID-19 testing decisions and behaviors. This study will focus on understanding factors associated with rapid COVID-19 testing, specifically. The primary objectives of the embedded study are to 1) Determine the effectiveness of community-level intervention using door-to-door recruitment and education in increasing COVID-19 testing and 2) Compare the effectiveness of the CHW- Facilitated Self-Sampling Intervention (FSSI) vs. CHW Testing Navigation Intervention (TNI).

DETAILED DESCRIPTION:
The pandemic landscape and people's experiences with testing, infection, and vaccination have changed dramatically over the past two years. Vaccines have become available, testing access in local communities has waxed and waned, and attitudes toward COVID-19 severity and susceptibility have shifted. Navigating the testing-decision landscape is confusing to the public (test availability for free versus charged or requiring insurance; testing and vaccination locations change; PCR versus antigen testing; home tests versus clinically delivered; symptom-based testing, exposure-driven testing, serial testing, resources to trust or not trust, etc.).

This study, referred to as the embedded study, builds off a broader population-based group randomized controlled trial (RCT) to evaluate the effects of a Facilitated Self-Sampling Intervention and Testing Navigation Intervention on testing behaviors. The embedded study will randomly select and assign priority block groups from the RCT to one of three arms - FSSI (n=16), TNI (n=16), or Control (n= 32). The allocation will be at a 2:1:1 rate across the three regions Houston/Harris County, South Texas, and Northeast Texas respectively. Community Health Workers will systematically sample and recruit 20 individuals from each PBG using a random start procedure. Study participants in the intervention arms will be enrolled, complete a baseline survey, receive a brief educational intervention, and complete a follow-up survey. Participants in the control arm will complete a baseline and follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older

Exclusion Criteria:

* Having been diagnosed with COVID-19 in the past 30 days based on a positive test (antigen or PCR) or a clinical diagnosis
* Having tested for COVID-19 with PCR or antigen test within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1232 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Testing completion by each study arm | between baseline and 2 months after the intervention
  Percent of participants from each study arm who complete testing (antigen or PCR)

SECONDARY OUTCOMES:
Number of participants who appropriately used antigen test as assessed by survey | baseline
  Appropriate use of antigen test is defined as taking the test when a test should have been taken (that is, symptoms present, known exposure to COVID).
Number of participants who appropriately used antigen test as assessed by survey | 2 months after the intervention
  Appropriate use of antigen test is defined as taking the test when a test should have been taken (that is, symptoms present, known exposure to COVID).
Number of participants with a positive test who took mitigation measures as assessed by survey | baseline
  Mitigation measures include mask wearing, isolating and notifying close contacts.
Number of participants with a positive test who took mitigation measures as assessed by survey | 2 months after the intervention
  Mitigation measures include mask wearing, isolating and notifying close contacts.
Number of participants who share antigen tests with close contacts who need to test as assessed by survey | baseline, 2 months after the intervention
Number of participants who share antigen tests with close contacts who need to test as assessed by survey | baseline
  Testing is needed for those with symptoms or known exposure to COVID.
Number of participants who share antigen tests with close contacts who need to test as assessed by survey | 2 months after the intervention
  Testing is needed for those with symptoms or known exposure to COVID.

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Fernandez, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Belinda M Reininger, DrPh, Principal Investigator — The University of Texas Health Science Center, Brownsville; David D McPherson, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Paul McGaha, DO, Principal Investigator — The University of Texas Health Science Center, Tyler; Marcia C de Oliveira Otto, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Kayo Fujimoto, PhD, Principal Investigator — The University of Health Science Center, Houston
Locations (3):
- United States (3):
  - The University of Texas Health Science Center, Brownsville, Brownsville, Texas
  - The University of Texas Health Science Center, Houston, Houston, Texas
  - University of Texas Health Science Center,Tyler, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No